CLINICAL TRIAL: NCT06334952
Title: Model-based Multichannel Transcranial Direct Current Electrical Stimulation (tDCS) in Drug-resistant Epilepsy: A Cross-over Study of Efficacy
Brief Title: Efficacy of Personnalized Transcranial Direct Current Electrical Stimulation (tDCS) in Drug-resistant Epileptic
Acronym: GALVANI GS-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: CRMBM-CEMEREM (Unknown); Institut National de la Santé Et de la Recherche Médicale, France - LTSI (Unknown); Neuroelectrics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RCAPHM23_0074; ID-RCB (Other: 2023-A02482-43)
Record Dates: First submitted 2024-03-16; First posted 2024-03-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy; Drug Resistant Epilepsy
Keywords: epilepsy; transcranial direct current stimulation; numerical models; quality of life
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Transcranial Direct Current Stimulation; Electroencephalography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS - Sham (Other): Patient will be randomized to firstly receive tDCS (10 non consecutive days, 20 minutes twice a day with 20 minutes of break) and then Sham (10 non consecutive days, 20 minutes twice a day with 20 minutes of break).
  Interventions: Device: transcranial direct current stimulation
- Sham - tDCS (Other): Patient will be randomized to firstly receive Sham (10 non consecutive days, 20 minutes twice a day with 20 minutes of break) and then tDCS (10 non consecutive days, 20 minutes twice a day with 20 minutes of break).
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Research MRI includes 3D-T1 weighted MRI (3D-T1), diffusion MRI (dMRI), resting-state functional MRI (rsfMRI).
  Other Names: Research MRI, EEG

SUMMARY:
The goal of this clinical trial is to to obtain a significant decrease in seizure frequency in patients with refractory focal epilepsy after applying treatment of cathodal tDCS, compared to sham stimulation drug-resistant epileptic patient. The main questions it aims to answer are:

* Changes in quality of life
* Percent of newly reported side effects after the stimulation period
* Scores in epilepsy severity. Participants will be randomized in a cross-over, and will receive 10 days of tDCS or Sham. Each day will allow 2 periods of 20 minutes stimulation separated by 20 minutes off (with 40 minutes of cathodal stimulation total).

ELIGIBILITY:
Inclusion Criteria:

1. Patient, parents or legal representative who have given written informed consent;
2. Age: ≥ 9 years;
3. Patients with drug-resistant focal epilepsy with no evolutive brain lesion and no surgical indication or with a previous surgical failure, refusing surgery or with a planned surgery compatible with the total duration of this study;
4. SEEG previously performed before inclusion with an adequate definition of the epileptogenic zone with all data required (pre-SEEG MRI, CT-scan or MRI with electrodes during SEEG and SEEG files) for personalization ;
5. Patient having a pre-SEEG 3D-T1 MRI and CT-scan with electrodes during SEEG available; This MRI can be done specifically for this trial or might be reused from EPINOV or NEURO7T trial)
6. For patients with VNS, experiencing no response or partial response, and for whom the stimulation parameters have been stable for at least 6 months
7. A research MRI scan that is suitable for navigated brain stimulation (NBS) and generation of electrical fields including dMRI for tractography;
8. Number of seizures ≥3/month during the baseline (before the first session of tDCS treatment);
9. Patient having stable medications for epilepsy 4 weeks before the baseline (except rescue treatment);
10. Patient's IQ, which in the investigator's opinion will enable questionnaires and neuropsychological assessments to be carried out;
11. Patient able to understand, speak and write in French;
12. Patient able to follow study's procedure;
13. Patient beneficiary or affiliated to a health insurance plan.

Exclusion Criteria:

1. Patients with seizures of generalized onset in the last 12 months;
2. Patient with multifocal epileptogenic zones, bilateral epileptogenic zone, or poorly defined epileptogenic zone. The epileptogenic network should not be restricted to the orbito frontal cortex or cingulate cortex;
3. Patients with psychogenic nonepileptic seizures;
4. Patient presenting a contraindication to MRI 3T (patient having a pacemaker, metallic foreign bodies, non-removably implanted electronic medical devices, claustrophobia, inability to remain in supine position, vagus nerve stimulator even when switched off is a contraindication for MRI 3T. EPINOV or NEURO 7T trial patients, who have accepted for their data to be reused, can be included even while wearing a VNS device) ;
5. Substance use abuse that may include alcohol , opioids (heroin, fentanyl) stimulants (Cocaine, methamphetamine) , hallucinogens (LSD, psilocybin (magic mushrooms), MDMA (Ecstasy))
6. Patient presenting a serious intercurrent pathology and/or a progressive brain tumor
7. Patient having damaged skin or scalp that may interfere with tDCS stimulation (e.g., eczema, lesion);
8. Patient having any cranial metal implants such as shrapnel or surgical clips (excluding <1 mm thick epicranial titanium skull plates and dental fillings) or medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant)
9. Patient having previous surgeries opening the skull leaving skull defects capable of allowing the insertion of a cylinder with a radius greater or equal to 5 mm;
10. Any condition that makes the study subject, in the opinion of the investigator, unsuitable for the study including presence of any disease, abnormality, medical or physical condition that, in the opinion of the investigator, may adversely impact, compromise, interfere, limit, affect or reduce the safety of the subject, the integrity of the data ;
11. Person protected by articles L1121-5, L1121-6 of Public Health Code (pregnant or breastfeeding woman, deprived of liberty by judicial decision, situations of social fragility, adults unable or unable to express their consent, person under judicial safeguard (article L1122-2)).

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2028-01-18 (Estimated)

PRIMARY OUTCOMES:
To obtain a significant seizure frequency change at the end of tDCS sessions compared to the seizure frequency calculated in the pre-treatment period of reference. | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Seizure frequency counting after end of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study.
To obtain a significant seizure frequency change at the end of tDCS sessions compared to the seizure frequency calculated in the pre-treatment period of reference. | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Seizure frequency counting after end of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study.
To obtain a significant seizure frequency change at the end of tDCS sessions compared to the seizure frequency calculated in the pre-treatment period of reference. | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Seizure frequency counting after end of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study.
To obtain a significant seizure frequency change at the end of tDCS sessions compared to the seizure frequency calculated in the pre-treatment period of reference. | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Seizure frequency counting after end of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study.

SECONDARY OUTCOMES:
Evaluation of the number of responders (defined as patient with >50% of seizure reduction) | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Proportion of responders evaluated after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluation of the number of responders (defined as patient with >50% of seizure reduction) | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Proportion of responders evaluated after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluation of the number of responders (defined as patient with >50% of seizure reduction) | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Proportion of responders evaluated after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluation of the number of responders (defined as patient with >50% of seizure reduction) | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Proportion of responders evaluated after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluate the number of seizure-free patients | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Number of seizure-free patients after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluate the number of seizure-free patients | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Number of seizure-free patients after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluate the number of seizure-free patients | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Number of seizure-free patients after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Evaluate the number of seizure-free patients | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Number of seizure-free patients after active session of 10 days of tDCS treatment compared to the baseline comparing Sham versus Active arms of the cross-over study
Quality of life after stimulation sessions with the baseline period | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Changes from baseline in the quality of life questionnaire (QOLIE 31 for adults and EFIQUACEE QOL for children) after the stimulation period
Quality of life after stimulation sessions with the baseline period | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Changes from baseline in the quality of life questionnaire (QOLIE 31 for adults and EFIQUACEE QOL for children) after the stimulation period
Quality of life after stimulation sessions with the baseline period | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Changes from baseline in the quality of life questionnaire (QOLIE 31 for adults and EFIQUACEE QOL for children) after the stimulation period
Quality of life after stimulation sessions with the baseline period | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Changes from baseline in the quality of life questionnaire (QOLIE 31 for adults and EFIQUACEE QOL for children) after the stimulation period
Evaluation of the change in seizure severity | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Changes in the scores of epilepsy severity (NHS3) (investigator evaluation)
Evaluation of the change in seizure severity | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Changes in the scores of epilepsy severity (NHS3) (investigator evaluation)
Evaluation of the change in seizure severity | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Changes in the scores of epilepsy severity (NHS3) (investigator evaluation)
Evaluation of the change in seizure severity | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Changes in the scores of epilepsy severity (NHS3) (investigator evaluation)
Changes in psychiatric comorbidities | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Changes from baseline in depression (NDDI-E) and anxiety (GAD-7) scores
Changes in psychiatric comorbidities | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Changes from baseline in depression (NDDI-E) and anxiety (GAD-7) scores
Changes in psychiatric comorbidities | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Changes from baseline in depression (NDDI-E) and anxiety (GAD-7) scores
Changes in psychiatric comorbidities | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Changes from baseline in depression (NDDI-E) and anxiety (GAD-7) scores
Safety assessment and possible side effects | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Percent of newly reported side-effect during and after the stimulation period
Safety assessment and possible side effects | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Percent of newly reported side-effect during and after the stimulation period
Safety assessment and possible side effects | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Percent of newly reported side-effect during and after the stimulation period
Safety assessment and possible side effects | V8 - 8 weeks after the end of the second cycle (each cycle is 10 days)
  Percent of newly reported side-effect during and after the stimulation period

OTHER OUTCOMES:
Compare brain functional connectivity before and after tDCS treatment | V5 - 8 weeks after the end of first cycle (each cycle is 10 days)
  Changes in functional connectivity measured by fMRI and EEG signal 4 weeks after the tDCS periods in comparison with baseline period
Evaluation of the impact of tDCS on interictal epileptic spikes (IESs) | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Change in the number of IESs per time unit after each tDCS session in comparison with baseline period
Evaluation of the impact of tDCS on interictal epileptic spikes | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Change in localization and extent of brain areas involved in IESs before and after each tDCS session in comparison with baseline period
Evaluation of the impact of tDCS on interictal epileptic spikes | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Change in localization and extent of brain areas involved in IESs before and after each tDCS session in comparison with baseline period
Evaluation of the impact of tDCS on interictal epileptic spikes | Visit 4 (V4) - 4 weeks after the end of first cycle (each cycle is 10 days)
  Changes in strength and density of functional links during IES before and after each tDCS session
Evaluation of the impact of tDCS on interictal epileptic spikes | V7 - 4 weeks after the end of the second cycle (each cycle is 10 days)
  Changes in strength and density of functional links during IES before and after each DCS session

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service de Neurophysiologie Clinique de l'Enfant et de L'Adulte, Pôle de Neurosciences Cliniques, Bordeaux
  - Département Neurologie Fonctionnelle et Epilepsie, Hôpital neurologique - Hospices Civils de Lyon, Bron
  - Service de Neurophysiologie clinique - Hôpital Roger Salengro, CHU Lille, Lille
  - Service Epileptologie et Rythmologie Cérébrale, Hôpital La Timone, Marseille
  - Service de Neurophysiologie clinique - GHU Psychiatrie et Neurosciences Sainte-Anne, Paris
  - Service de Neurologie - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Explorations neurophysiologiques - Pôle neurosciences, CHU de Toulouse, Hôpital Pierre Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No